CLINICAL TRIAL: NCT07016477
Title: Prospective Registry of Patients Undergoing Cardiac CT With NAEOTOM Alpha Photon Counting-detector CT Before Transcatheter Aortic Valve Implantation
Brief Title: Prospective Registry of Patients Undergoing Cardiac CT With NAEOTOM Alpha PCD-CT Before TAVI Procedure
Acronym: Alpha Registry
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Prof. Maurovich-Horvat Pál, PhD, MPH, DSc, Director of Medical Imaging Centre, Chairman of Radiology, Semmelweis University
Other Study IDs: BM/9095-1/2024
Record Dates: First submitted 2025-02-23; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Aortic Valve Stenosis; Tomography, X-Ray Computed
Keywords: photon-counting detector computed tomography
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Aortic stenosis: Patients with aortic valve disease for whom transcatheter aortic valve implantation is indicated and who present for pre-interventional evaluation will be enrolled after written consent.
  Interventions: Diagnostic Test: Ultra-High Resolution Photon Counting Detector Coronary Computed Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Ultra-High Resolution Photon Counting Detector Coronary Computed Tomography Angiography — Clinically indicated Ultra-High Resolution Photon-Counting Detector Coronary Computed Tomography Angiography (UHR PCD-CT CCTA) for the pre-procedural evaluation of patients scheduled to undergo transcatheter aortic valve implantation.
  Other Names: Photon-Counting Detector CT (Naeotom Alpha, Siemens Healthineers)

SUMMARY:
The clinical and demographic characteristics of patients undergoing transcatheter aortic valve implantation (TAVI) pose unique challenges for coronary computed tomography (CT) imaging, as this patient population is mainly composed of elderly, frail individuals with severe aortic stenosis, multiple comorbidities, high prevalence of heavily calcified coronary artery disease (CAD) and revascularized coronary arteries. Such vulnerable patients could benefit from a more precise assessment and characterization of their CAD with ultra-high resolution (UHR) photon-counting detector (PCD) CT that would potentially avoid the need for pre-implantation invasive coronary angiography (ICA). This international multicenter prospective registry study aims to investigate the feasibility and diagnostic accuracy of PCD-CT in the assessment of CAD in the high-risk population of patients undergoing TAVI, as compared to ICA.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated TAVI
* Clinically indicated CT and invasive coronary angiography
* There are no contraindications to CT angiography.
* Understanding and signing the consent form

Exclusion Criteria:

* Pregnancy or breastfeeding
* Chronic renal failure (eGFR <30 ml/m2)
* Active oncological treatment
* Any condition for which TAVI is contraindicated and therefore no prior radiological investigation of TAVI is indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with aortic valve stenosis for whom TAVI is indicated and who present for pre-operative investigation.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Ultra-High Resolution Photon-Counting Detector Coronary Computed Tomography Angiography (UHR PCD-CT CCTA) | through study completion, an average of 2 years
  Assessment of the diagnostic accuracy (sensitivity, specificity, PPV, NPV) of UHR PCD-CT coronary angiography as compared to invasive coronary angiography (ICA) within three months of PCD-CT

SECONDARY OUTCOMES:
Image Noise Analysis Across Reconstruction Parameters | through study completion, an average of 2 years
  Quantitative assessment of image noise (measured in HU) in CT images reconstructed with varying parameters, including reconstruction kernel type, quantum iterative reconstruction (QIR) levels, and slice thickness.
Correlation of Image Noise and Body Mass Index | through study completion, an average of 2 years
  Correlation of image noise (measured in HU) and body mass index (kg/m2) across different image reconstruction parameters, including kernel type, quantum iterative reconstruction (QIR) level, and slice thickness.
Correlation of Image Noise and Heart Rate | through study completion, an average of 2 years
  Correlation of image noise (measured in HU) and heart rate (bpm) across different image reconstruction parameters, including kernel type, quantum iterative reconstruction (QIR) level, and slice thickness.
Contrast-to-Noise Ratio (CNR) Analysis Across Reconstruction Parameters | through study completion, an average of 2 years
  Quantitative assessment of contrast-to-noise ratio (unitless) in CT images reconstructed with varying parameters, including reconstruction kernel type, quantum iterative reconstruction (QIR) levels, and slice thickness.
Vessel Sharpness Analysis Across Reconstruction Parameters | through study completion, an average of 2 years
  Quantitative assessment of vessel sharpness (measured in 1/mm) in CT images reconstructed with varying parameters, including reconstruction kernel type, quantum iterative reconstruction (QIR) levels, and slice thickness.
Blooming Analysis Across Reconstruction Parameters | through study completion, an average of 2 years
  Quantitative assessment of blooming (percentage) in CT images reconstructed with varying parameters, including reconstruction kernel type, quantum iterative reconstruction (QIR) levels, and slice thickness.
Subjective Image Quality Analysis | through study completion, an average of 2 years
  Overall image quality, image noise and vessel sharpness assessed on a 4-point Likert scale (1 = non-diagnostic, 4 = excellent) by 2 blinded readers/site. Comparison of image quality between reconstructions with varying parameters, including reconstruction kernel type, quantum iterative reconstruction (QIR) levels, and slice thickness.
Correlation of Quantitative Coronary Artery Disease Assessment | through study completion, an average of 2 years
  Correlation and agreement of percent diameter stenosis (PDS) measured on UHR PCD-CT dataset and quantitative coronary angiography (QCA).
Correlation of Quantitative In-Stent Restenosis Assessment | through study completion, an average of 2 years
  Correlation and agreement of quantitative in-stent restenosis (ISR) measured on UHR PCD-CT dataset and quantitative coronary angiography (QCA).
Correlation of Fractional Flow Reserve Measurement | through study completion, an average of 2 years
  Correlation and agreement of CT-based fractional flow reserve (FFR-CT) measured on UHR PCD-CT dataset and invasive fractional flow reserve.
Quantitative Assessment of Plaque Composition | through study completion, an average of 2 years
  Measure the volume of plaque components (in mm3) on UHR PCD-CT datasets across different image reconstruction parameters, including kernel type and quantum iterative reconstruction (QIR) level.
Correlation of Plaque Composition | through study completion, an average of 2 years
  Correlation and agreement of plaque composition assessment from UHR PCD-CT dataset and intracoronary techniques such as optical coherence tomography (OCT) in patients who had both tests done.
Quantitative Assessment of Extracellular Volume Fraction | through study completion, an average of 2 years
  Quantitative analysis of the extracellular volume (ECV) fraction measured on PCD-CT dataset.
Analysis of Structured Coronary Artery Disease Reporting in UHR PCD-CT | through study completion, an average of 2 years
  Analysis of coronary artery disease classification according to the Coronary Artery Disease-Reporting and Data System (CAD-RADS 2.0).
Correlation of Quantitative UHR PCD-CT CCTA Parameters with Ischemia Imaging Tests | through study completion, an average of 2 years
  Correlation of quantitative UHR PCD-CT CCTA parameters with the results of additional imaging ischemia tests in patients who had both PCD-CT CCTA and one of the following tests done: stress echocardiography, stress single photon emission computed tomography (SPECT), stress positron emission tomography (PET), and stress magnetic resonance imaging (MRI).
Correlation of Quantitative UHR PCD-CT CCTA Parameters with Other Imaging Tests | through study completion, an average of 2 years
  Correlation of quantitative UHR PCD-CT CCTA parameters with the results of additional imaging tests in patients who had both PCD-CCTA and one of the following tests done: transthoracic echocardiography, transesophageal echocardiography, cardiac MRI.
Correlation Between PCAT Attenuation and CT-derieved or Clinical Parameters | from inclusion up to a maximum follow-up period of 5 years
  To assess the correlation between pericoronary adipose tissue (PCAT) attenuation (measured in HU on UHR PCD-CT CCTA data) and (1) anatomical severity of CAD (percent diameter stenosis), (2) functional severity of disease (FFR-CT), (3) plaque composition and (4) clinical outcome.
Correlation Between EAT Attenuation and CT-derieved or Clinical Parameters | from inclusion up to a maximum follow-up period of 5 years
  To assess the correlation between epicardial adipose tissue (EAT) attenuation (measured in HU on UHR PCD-CT CCTA data) and (1) anatomical severity of CAD (percent diameter stenosis), (2) functional severity of disease (FFR-CT), (3) plaque composition and (4) clinical outcome.
Lung Water Density Quantification | through study completion, an average of 2 years
  Measurement of lung water density by virtual non-contrast CT and iodine mapping CT, compared to non-contrast CT.
Assessment of Whole Body Extracellular Volume | through study completion, an average of 2 years
  Assessment of whole body extracellular volume (ECV) in patients undergoing TAVI compared to healthy volunteer controls scanned in a separate study.
Major Adverse Cardiac Events | from inclusion up to a maximum follow-up period of 5 years
  Composite endpoint of major adverse cardiovascular event (MACE); defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, stroke.
Extended Major Adverse Cardiovascular Events | from inclusion up to a maximum follow-up period of 5 years
  Composite endpoint of major adverse cardiovascular event (MACE); defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, stroke, unstable angina, or heart failure admission
Prosthesis Function Evaluation | from inclusion up to a maximum follow-up period of 5 years
  Subjective analysis of prosthesis function using UHR and spectral PCD-CT data to detect pathologies e.g. hypoattenuating leaflet thickening (HALT).
Cost-effectiveness | from inclusion up to a maximum follow-up period of 5 years
  Costs of PCD-CT and complications compared with costs of ICA and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Pál Maurovich-Horvat, MD, PhD, DSc, Principal Investigator — Semmelweis University
Locations (7):
- Medical University of South Carolina, Charleston, South Carolina, United States
- Germany (3):
  - Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau
  - University Medical Center Mainz, Mainz
  - Universitätsklinikum Tübingen, Tübingen
- Semmelweis University, Budapest, Hungary
- Maastricht University, Maastricht, Netherlands
- University Hospital of Zürich, Zurich, Switzerland